CLINICAL TRIAL: NCT02573415
Title: Uterine Transplantation for the Treatment of Uterine Factor Infertility
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Michelle Kuznicki, Staff Physician, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLA 14-085
Record Dates: First submitted 2015-10-08; First posted 2015-10-09 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Primary Uterine Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Uterus Transplantation (Experimental): Women will undergo deceased donor uterine transplantation after IVF.
  Interventions: Procedure: Uterus Transplant

INTERVENTIONS:
Procedure: Uterus Transplant — transplant of a deceased donor uterus.

SUMMARY:
This feasibility study aims to enroll ten subjects who will undergo deceased donor uterine transplantation at Cleveland Clinic. We estimate that fifty to one hundred patients with uterine factor infertility will need to be screened to identify 10 appropriate subjects.

There are seven phases involved in this study: Primary and Secondary Screening, Medical Evaluation, IVF, Transplantation, Embryo Transfer, Pregnancy/Delivery and Follow up

DETAILED DESCRIPTION:
Uterine factor infertility (UFI) is one of the few irreversible causes of female infertility. Until recently, no medical or surgical options have been available for women with this diagnosis. UFI is defined by the lack of a functional uterus; this condition can either be congenital (e.g. Rokitansky syndrome, where a woman is born without an intact uterus) or acquired (e.g. resulting from hysterectomy or damage to the uterus from procedures or infections).

Uterine infertility affects 3-5% of the female population. It is estimated that there are at least 50,000 women of reproductive age with uterine infertility in the United States. Existing options for women affected by UFI are limited to adoption or maternal surrogacy. Surrogacy involves harvesting eggs from the UFI patient and fertilizing these eggs in a lab with the intention of implanting fertilized embryos into a third party who will carry the pregnancy. Adoption and surrogacy are considered acceptable options for many women with UFI. For others, due to social, ethical, cultural and/or religious reasons, these options are not permissible. In many countries around the world, maternal surrogacy is illegal, leaving no option for UFI patients to conceive a biological child.

Recently, uterine transplantation has been proposed as an alternative method of treating UFI. Uterine transplantation is intended as a life enhancing procedure, not a life saving procedure, and is considered to be similar to transplants of the face, extremities and pancreas. Interestingly, uterine transplantation is considered an "ephemeral" transplant, and is not intended to last for the duration of the life of the recipient. The transplant is maintained for only as long as is necessary to produce one or two offspring for the patient.

The need for novel approaches to UFI is clear and exciting work from a team of investigators in Sweden has finally demonstrated this year that uterine transplantation can result in the successful delivery of healthy infants with minimal risk to the mother. After careful collaboration with this Swedish group, we now aim to bring the first uterine transplantation protocol to the United States using a multidisciplinary team of investigators from within the Cleveland Clinic.

There have been 11 uterine transplants performed in humans worldwide. The first uterine transplant was performed in Saudi Arabia in 2000. The living-donor graft survived for 3 months and was subsequently removed due to graft failure. The failure of the graft was attributed to thrombosis (blood clots affecting the circulation to the organ). Pregnancy was never attempted using the transplanted uterus prior to it being removed.

This year, Brännström M. et al. published their experience with the first clinical trial of human uterine transplantation in a series of 9 women. The clinical trial, based in Sweden, began in 2012 under Institutional Review Board (IRB) approval from the University of Gothenburg. The nine women in the study group received uteri from living donors and the report, published in Fertility and Sterility in May 2014, described that seven out of the nine transplants were viable after six months of follow up. Nonviability of the two grafts was reportedly due to uterine artery thrombosis. In most cases, donors were the recipient's mother. Eight of the recipients had Rokitansky syndrome. One recipient had undergone a hysterectomy for cervical cancer. There were no immediate perioperative complications and all patients with successful grafts began to have spontaneous menstrual periods within a few months of transplantation. Mild rejection appeared to be treatable with steroids. All recipients had 10 viable embryos produced by in vitro fertilization performed prior to uterine transplantation. Those embryos were then transferred into the transplanted uterus to achieve pregnancy. This research has now resulted in the first published report of a human live birth from uterine transplantation.

In the Gothenburg experience, the donor operation consisted of a hysterectomy including the uterine arteries and veins with the branches of the internal iliac artery and vein and vault of vagina. The first segment of the ovarian veins caudad to the ovaries (in order to protect their outflow) was also included. The explanted uterus was perfused with chilled University of Wisconsin (UW) solution and prepared for implantation. The implantation was achieved by anastomosis into the iliac vessels bilaterally, in some cases the donor ovarian veins where included. The vault of the donor vagina was anastomosed into the existing vagina or neovagina. Immunosuppression following uterine transplantation included induction with thymoglobulin and maintenance with tacrolimus, mycophenolate mofetil and oral steroids. Mycophenolate mofetil was discontinued before pregnancy attempts as it is contraindicated in pregnancy. This immunosuppression regimen is similar to the regimen proven effective in kidney transplantation, another solid organ graft.

Dr. Andreas Tzakis has been working closely with the Gothenburg group through both early animal models as well as the recent clinical trial in humans. Below is a summary of this group's published relevant findings:

1. Two grafts were lost (one soon after transplant and the other 4 months later) due to uterine artery thrombosis.
2. One donor had a surgical complication, her ureter was injured during removal of the uterus, and she required a late ureteral reimplantation due to ischemic damage of her ureter
3. Five recipients developed mild rejection of the graft. This was detected by cervical biopsy and was treated successfully with steroids in all cases.
4. Menstruation occurred regularly in all seven subjects with a successful transplant within a few months of transplantation.
5. One documented subject had one live birth by Cesarean section; this pregnancy was complicated by preeclampsia (high blood pressure of pregnancy) at 31.5 weeks gestation

4. Pregnancy after Solid Organ Transplantation

Since only one live birth in human uterine transplant recipients has been reported, the pregnancy risks are not firmly established; however pregnancies and deliveries after uterine transplantation of healthy offspring have been accomplished in small and large animals (mice, rats, sheep, nonhuman primates). In addition, pregnancy after other solid organ transplants in humans is well documented.

The use of immunosuppressive medication is well studied in pregnancy after solid organ transplantation as well as in women with certain rheumatologic conditions and inflammatory bowel disease. Tacrolimus and cyclosporine are among the most widely used in pregnancy. Birth defects with cyclosporine or tacrolimus occur at an incidence of 4-5% which is no different than the general population. Cyclosporine is associated with low birth weight but does not appear to impact long term outcomes including intelligence quotient (IQ). Mycophenolate mofetil (MMF) is associated with a specific pattern of birth defects including facial malformations, finger abnormalities and heart defects. This medication should not be used in the first trimester of pregnancy. Azathioprine does not cause birth defects. Corticosteroids are considered safe however high doses can increase the risk of premature rupture of membranes. Immunosuppression is also noticed in infants exposed to these medications during pregnancy including low immunoglobulin levels and lymphocyte counts. Most of these deficits seem to normalize by the sixth month of life, with no noted impact on the infants' health.

Renal transplant is the most common solid organ transplant after which pregnancy has been reported. In these women over 90% achieve successful pregnancy outcomes after the first trimester. Pregnancy risks include low birth weight, preterm delivery and preeclampsia. It has consistently been shown that pregnancy does not adversely affect the graft function or survival.

The most frequent maternal complication in this patient population is pregnancy induced hypertension. Management of such pregnancy complications uterine transplant recipients should follow standard obstetric guidelines.

Prematurity is the main fetal complication, which affects nearly 40% of live births. The mean reported gestational age at delivery is 36.5 weeks, while the mean birth weight is approximately 14% less than general population (6 lb 5 oz vs 7 lb 4 oz). Other fetal complications that have been observed include intrauterine growth restriction (approximately 20%), prenatal infections, and birth defects.

Over 400 pregnancies after liver transplantation have been reported. Similar risks are reported in these women including preeclampsia preterm birth and low birth weight. Less data is available from women who have undergone less common transplants. Kidney-pancreas transplant is associated with a higher complication rates. Hypertension is reported and 75% in addition there is a 55% risk of infection and 68% risk of low birth weight. These studies are limited by lack of consideration of the original disease of the organ recipient or the functional status of the transplanted organ. Women undergoing uterine transplantation will have no significant preexisting medical conditions unlike women undergoing other solid organ transplantations. Both these elements are likely to have an influence on the incidence of complications of the pregnancy and have not been included in previous large analyses.

According to The American Society of Transplantation, pregnancy is allowable in renal organ transplantation one year after transplantation if there has been no signs of rejection, the transplanted organ has adequate function, there is no active infection (particularly cytomegalovirus infection) and the immunosuppression dose has been stable.

Waiting one year after the transplantation prior to conception decreases the risk of acute rejection and infection. During the pregnancy it is important to monitor blood pressure and treat hypertension diligently, maintain strict glycemic control, monitor for signs of infection, and assess maternal levels of immunosuppressive medications more frequently.

ELIGIBILITY:
Inclusion Criteria:

1. Must meet criteria for uterine factor infertility

   1. Prior hysterectomy
   2. Congenital absence or malformation of the uterus preventing pregnancy c, Infertility due to uterine damage from prior injury or infection
2. Must be between the ages of 21-45 and the embryos must have been produced between the age of 21-39. (age at the time the embryos are produced, not current age)
3. Must be willing to undergo a psychiatric and social work pre-transplant evaluation
4. Must be willing to undergo general anesthesia, in vitro fertilization, major gynecologic surgery, pregnancy with potential high risk complications, cesarean delivery and eventual hysterectomy to remove the graft
5. Must be willing and able to receive potent immunosuppressive medications and must be able to follow standard infection prophylaxis protocols
6. Must be willing to receive standard vaccinations such as influenza, pneumococcus, human papillomavirus (HPV) and hepatitis B
7. Must be willing and able to sign informed consent and follow all outlined procedures and recommendations in the protocol

Exclusion Criteria:

1. History of hypertension, diabetes, or significant heart, liver, kidney or central nervous system disease
2. Any medical diagnosis placing the subject at high risk of surgical complications based on the transplant team's review of medical history.
3. Current smoker (smoking cessation must have occurred 3 months prior to enrollment)
4. History of prior malignancy except for cervical cancer in stage 1a or 1b after 3 years.
5. Human immunodeficiency virus, mycobacteria, hepatitis B (Hepatitis risk is for those with hepatitis B (HB) surface and/or core antigen and/or hepatitis B virus (HBV) DNA positive. Thos that are HB core antibody positive are at minimal risk and everyone else is not at risk), or hepatitis C.
6. Presence of active documented systemic infection or recent systemic infection within the past three months
7. Chemical and/or alcohol dependency or abuse
8. Presence of low lying pelvic kidney(s). Pelvic and horse shoe kidneys are common in the Rokitansky syndrome, and occur with a frequency as high as 30-40%. These abnormalities are usually known to subjects as part of their Mullerian agenesis diagnosis. If the patient is unsure about the status of their kidneys, the performance of a renal ultrasound is considered standard of care. These patients need to be informed of any kidney abnormalities, as they are frequently associated with kidney stones or obstructive kidney disease.
9. BMI greater than 30 kg/m2

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-10; Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of successful live births after uterus transplant and IVF | 2 years after transplantation
  Full term birth by cesarian section after IVF followed by uterus transplant

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Kuznicki, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Johannesson L, Humphries LA, Porrett PM, Testa G, Anderson S, Walter JR, Rush M, Ferrando CA, O'Neill K, Richards EG. Classification and treatment of vaginal strictures at the donor-recipient anastomosis after uterus transplant. Fertil Steril. 2024 Sep;122(3):525-534. doi: 10.1016/j.fertnstert.2024.04.019. Epub 2024 Apr 16. PMID 38636770
- [Derived] Walter JR, Johannesson L, Falcone T, Putnam JM, Testa G, Richards EG, O'Neill KE. In vitro fertilization practice in patients with absolute uterine factor undergoing uterus transplant in the United States. Fertil Steril. 2024 Sep;122(3):397-405. doi: 10.1016/j.fertnstert.2024.04.017. Epub 2024 Apr 15. PMID 38631504
- [Derived] Richards EG, Agatisa PK, Davis AC, Flyckt R, Mabel H, Falcone T, Tzakis A, Farrell RM. Framing the diagnosis and treatment of absolute uterine factor infertility: Insights from in-depth interviews with uterus transplant trial participants. AJOB Empir Bioeth. 2019 Jan-Mar;10(1):23-35. doi: 10.1080/23294515.2019.1572672. Epub 2019 Mar 11. PMID 30855220
- [Derived] Arian SE, Flyckt RL, Farrell RM, Falcone T, Tzakis AG. Characterizing women with interest in uterine transplant clinical trials in the United States: who seeks information on this experimental treatment? Am J Obstet Gynecol. 2017 Feb;216(2):190-191. doi: 10.1016/j.ajog.2016.11.1028. Epub 2016 Nov 16. No abstract available. PMID 27865979